CLINICAL TRIAL: NCT04180631
Title: Diagnostic Value of Quantitative Ultrasound Imaging Parameters for Hepatic Steatosis in Patients With Non-alcoholic Fatty Liver Disease
Brief Title: Quantitative US for Hepatic Steatosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Samsung Medison (Industry)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SNUH-1808-155-967
Record Dates: First submitted 2019-01-08; First posted 2019-11-27 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Hepatic Steatosis
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quantitative ultrasound imaging parameter (Experimental): Quantitative ultrasound imaging parameter (QUS)
  Interventions: Diagnostic Test: Quantitative ultrasound imaging parameter (QUS)

INTERVENTIONS:
Diagnostic Test: Quantitative ultrasound imaging parameter (QUS) — Quantitative ultrasound imaging parameters (QUS) are analyzed to evaluate hepatic steatosis

SUMMARY:
The purpose of this study is to investigate the diagnostic performance of quantitative ultrasound imaging parameter for the assessment of hepatic steatosis in patients with non-alcoholic fatty liver disease using magnetic resonance imaging proton density fat fraction (MRI-PDFF) and MR spectroscopy as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* patients with clinically suspected non-alcoholic fatty liver disease (NAFLD) or non-alcoholic steatohepatitis (NASH), or living-donor candidates for liver transplantation, or volunteers
* Signed informed consent

Exclusion Criteria:

* chronic liver disease patients (serum HBsAg positive or anti-hepatitis C virus (HCV), histologic confirmation)
* chronic alcoholics
* serum alanine transaminase (ALT)>5 times the upper limit of normal within 3 months
* previous liver surgery
* acute hepatitis or bile duct obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2020-01-19 (Actual); Study Completion 2020-01-19 (Actual)

PRIMARY OUTCOMES:
Correlation between quantitative US imaging parameter (QUS) and MR fat fraction | 3 months
  reference standard: MR spectroscopy or MRI-proton density fat fraction value

SECONDARY OUTCOMES:
Diagnostic performance of QUS to detect mild fatty liver and moderate fatty liver | 3 months
  reference standard: MR fat fraction
Correlation between S-shearwave elastography and MR elastography | 3 months
  Reference standard: liver stiffness at MR elastography, using Pearson's correlation analysis or Spearman rank correlation analysis
Intra-observer agreement of quantitative ultrasound imaging parameter | same 1 day
  intraclass correlation coefficient (ICC)
Development and validation of deep learning model for prediction of hepatic steatosis | 1 month
  ROC analysis and C-index for deep learning model for prediction of hepatic steatosis

CONTACTS AND LOCATIONS:
Overall Officials: Jeon Min Lee, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jeon SK, Lee JM, Joo I, Yoon JH, Lee G. Two-dimensional Convolutional Neural Network Using Quantitative US for Noninvasive Assessment of Hepatic Steatosis in NAFLD. Radiology. 2023 Apr;307(1):e221510. doi: 10.1148/radiol.221510. Epub 2023 Jan 3. PMID 36594835